CLINICAL TRIAL: NCT07151937
Title: A Seamless Phase 2a/2b, Randomized, Double-Blind, Placebo- and Active-Controlled, Multiple-Arm, Multiple-Stage, Adaptive Study Evaluating the Efficacy and Safety of LAD191 in Adults With Moderate-to-Severe Hidradenitis Suppurativa
Brief Title: A Study of LAD191 in Adults With Hidradenitis Suppurativa
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-27134-10; 2025-521293-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-02; First posted 2025-09-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: A double-blind, multiple-arm, adaptive treatment-selection designed study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- LAD191 Dose A (Experimental): Participants will receive dose A LAD191 subcutaneous (SC) injection during both Treatment Period 1 and Treatment Period 2, unless if Dose A is eliminated after interim analysis, participants will receive the highest available dose of LAD191 during Treatment Period 2.
  Interventions: Drug: LAD191
- LAD191 Dose B (Experimental): Participants will receive dose B LAD191 SC injection during both Treatment Period 1 and Treatment Period 2, unless if Dose B is eliminated after interim analysis, participants will receive the highest available dose of LAD191 during Treatment Period 2.
  Interventions: Drug: LAD191
- LAD191 Dose C (Experimental): Participants will receive dose C LAD191 SC injection during both Treatment Period 1 and Treatment Period 2, unless if Dose C is eliminated after interim analysis, participants will receive the highest available dose of LAD191 during Treatment Period 2.
  Interventions: Drug: LAD191
- Placebo (Placebo Comparator): Participants will receive matching LAD191 placebo SC injection during Treatment Period 1 and will begin treatment with the highest available dose of LAD191 during Treatment Period 2.
  Interventions: Drug: LAD191; Other: Placebo
- Adalimumab (Active Comparator): Participants will receive adalimumab SC injection during Treatment Period 1 and will begin treatment with the highest available dose of LAD191 during Treatment Period 2.
  Interventions: Drug: LAD191; Drug: Adalimumab

INTERVENTIONS:
Drug: LAD191 — LAD191 subcutaneous injection.
Other: Placebo — LAD191 Placebo subcutaneous injection.
  Arms: Placebo
Drug: Adalimumab — Adalimumab subcutaneous injection.
  Arms: Adalimumab

SUMMARY:
The main purpose of this study is to assess the efficacy of multiple dosing regimens of LAD191 compared to placebo in participants with moderate-to-severe Hidradenitis Suppurativa (HS) and to access the safety, tolerability, pharmacokinetic and immunogenicity in participants with moderate-to-severe HS.

DETAILED DESCRIPTION:
The purpose of this study is to assess the multiple dosing regimens of LAD191 compared to placebo in participants with moderate-to-severe Hidradenitis Suppurativa (HS). The study has a prospectively defined adaptive design that will utilize interim data for futility evaluation.

The study includes up to 4 weeks screening period 16-week double-blind, placebo-controlled period (Treatment period 1), 16-weeks LAD191 double-blind period (Treatment period 2), and 12-week safety follow-up.

The study participants will be randomized to one of the following treatment arms: LAD191 dose A, LAD191 dose B; LAD191 dose C, Adalimumab or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to (>=) 18 to less than or equal to (<=) 65 years.
* A diagnosis of moderate-to-severe HS defined as a total of >= 5 inflammatory lesions (i.e., number of abscesses plus number of inflammatory nodules) at both the Screening and Baseline/Day 1 visits, with signs and symptoms of HS for at least 6 months.
* HS lesions present in at least 2 distinct anatomic areas (e.g., left and right axilla), one of which must be at least Hurley Stage II or Hurley Stage III at both the Screening and Baseline/Day 1 visits.
* History of inadequate response, intolerance, or contraindication to a course of a systemic antibiotics for treatment of HS at the screening visit.
* Regular use of over-the-counter topical antiseptics on HS lesions and agrees to regular use, throughout the entirety of the study.
* Participants who are women of child-bearing potential (WOBCP) and male participants must agree to the requirements for the avoidance of pregnancy and exposure of the participant's partner to LAD191 during the study.

Exclusion Criteria:

* HS with >20 draining tunnels at the Screening or Baseline/Day 1 visit.
* Ongoing medical conditions requiring systemic immunosuppressive/immunomodulating treatments during the study.
* Known hypersensitivity to LAD191 or any of its excipients.
* Known hypersensitivity to adalimumab or biosimilar or any of its excipients or meeting any warning or contraindication to adalimumab treatment as per the approved product information, and as per the Investigator's judgment.
* Hypersensitivity or systemic reaction to a prior biologic (antibody-based) therapy, regardless of indication, that was clinically significant, as per the Investigator's judgment.
* Prior treatment with LAD191.
* Live or attenuated vaccinations 4 weeks prior to Baseline/Day 1 or is planning to receive any such vaccine during the study.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
* Intention to use any concomitant medication or therapy that is not permitted by this protocol or failure to meet the required washout period for a particular prohibited medication prior to Baseline/Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving 50 Percent (%) Reduction from Baseline in Hidradenitis Suppurativa Clinical Response (HiSCR-50) | At Week 16
  HiSCR-50 is defined as ≥50% reduction in total AN count, with no increase in abscess count, and no increase in draining fistula count relative to baseline.

SECONDARY OUTCOMES:
Proportion of Participants Achieving 75% Reduction from Baseline in HiSCR-75 at Week 16 | At Week 16
  HiSCR-75 is defined as ≥75% reduction in total AN count, with no increase in abscess count, and no increase in draining fistula count relative to baseline.
Proportion of Participants Achieving 90% Reduction from Baseline in HiSCR-90 at Week 16 | At Week 16
  HiSCR-90 is defined as 90% reduction in total AN count, with no increase in abscess count, and no increase in draining fistula count relative to baseline.
Proportion of Participants Achieving 55% Reduction from Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4-55) at Week 16 | At Week 16
  The IHS4 is determined by counting nodules, abscesses, and draining tunnels (fistulae/sinuses). IHS4 (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or lower indicates a mild stage of hidradenitis suppurativa, a score of 4-10 indicates a moderate stage, and a score of 11 or higher indicates a severe stage of the disease. IHS4-55, is a dichotomous IHS4 variable based on a ≥55% reduction of the total score.
Change from Baseline in Skin Pain Numerical Rating Scale (NRS) at Week 16 | At Week 16
  Skin Pain NRS is an 11-point scale in which patients are asked to rate their skin pain over the prior 24 hours, where 0 is no skin pain and 10 is pain as bad.
Change from Baseline in Hidradenitis Suppurativa Quality of Life (HiSQOL) at Week 16 | At Week 16
  The HiSQOL was specifically developed for use in clinical trials to assess Quality of Life (QoL) and comprises a 17-item questionnaire grouped into 3 sub-scales covering symptoms, psychosocial, and activity-adaptation aspects, with a recall period of seven days. Each item is structured as a Likert-type scale with five or seven response levels and, for all items, the score ranges from 0 (not at all) to 4 (extremely). Individual item scores are summed and a total score ranging from 0 to 68 is calculated, where the higher the score the more impact HS has on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.

IPD SHARING:
Plan to Share IPD: No